CLINICAL TRIAL: NCT01238770
Title: A Phase I/II Study of Pazopanib (GW786034) and Cyclophosphamide in Patients With Platinum-resistant Recurrent, Pre-treated Ovarian Cancer
Brief Title: Phase I/II Study of Pazopanib and Cyclophosphamide in Patients With Platinum-resistant Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Priv.-Doz. Dr. med. Joachim Rom (Other)
Responsible Party: Sponsor-Investigator, Priv.-Doz. Dr. med. Joachim Rom, PD Dr. med, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3107000
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — pazopanib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamid + Pazopanib (Experimental): Cyclophosphamid + Pazopanib
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Phase I Cyclophosphamid Pazopanib Dose level I 50 mg/day 400 mg/day Dose level II 50 mg/day 600 mg/day Dose level III 50 mg/day 800 mg/day
  Cyclophosphamide 50 mg daily orally Pazopanib 400, 600 or 800 mg daily orally
  Phase II:
  Cyclophosphamide 50 mg daily orally Pazopanib 400, 600 or 800 mg daily orally The dose for the phase II part of the trial will be based on the MTD of phase I.
  Other Names: Cyclophosphamid

SUMMARY:
The current trial shall clarify the potential of the multitarget antiangiogenic tyrosinkinase inhibitor GW 786034 (pazopanib) in combination with oral cyclophosphamide as salvage treatment in patients with recurrent, pretreated ovarian cancer.

DETAILED DESCRIPTION:
This study is a prospective open-label, non-randomized multicenter phase I/II trial in order to determine overall response rate of patients with platinum-resistant or refractory recurrent, pretreated epithelial ovarian cancer.

In order to assure adequate toxicity assessment, a phase-I-trial is proponed. Phase II will be performed with MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Female subjects ≥18 years of age
3. Histologically or cytologically confirmed diagnosis of: epithelial ovarian cancer which is platinum resistant or platinum refractory,cancer of the fallopian tube, peritoneal cancer
4. Patients must have failed available standard chemotherapy regimen
5. Prior treatment with at least 2 chemotherapy regimens in advanced tumor setting
6. Performance status ECOG 0 - 2
7. Adequate contraception
8. Adequate organ function
9. Measurable disease according to RECIST criteria.
10. Able to swallow and retain oral medication.
11. Life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Any second malignancy within the last 5 years, with the exception of basal cell or squamous cell skin cancer or in situ carcinoma of the cervix uteri
2. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug.
3. Clinically significant gastrointestinal abnormalities which might interfere with oral dosing
4. Any unstable or serious concurrent condition (e.g., active infection requiring systemic therapy).
5. Prolongation of corrected QT interval (QTc) >480 msecs.
6. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Symptomatic peripheral vascular disease
   * Coronary artery by-pass graft surgery
   * Class II, III or IV congestive heart failure as defined by the New York Heart Association (NYHA)
   * History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
7. Macroscopic hematuria
8. Hemoptysis that is clinically relevant within 4 weeks of first dose of study drug
9. Evidence of active bleeding or bleeding diathesis
10. Known endobronchial lesions or involvement of large pulmonary vessels by tumor
11. Prior major surgery or trauma within 14 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
12. Chemotherapy or radiation therapy within 2 weeks prior to the first dose of study drug.
13. Biological therapy, hormonal therapy or treatment with an investigational agent within 28 days or 5 half-lives
14. Prior antiangiogenic therapy.
15. Is unable or unwilling to discontinue predefined prohibited medications listed in the protocol for 14 days or five half-lives of a drug (whichever is longer) prior to Visit 1 and for the duration of the study
16. Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity.
17. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib
18. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
19. Pregnancy
20. More than 3 different chemotherapy regimens in advanced tumor setting
21. Uncontrolled hypertension
22. History of ischemic event (stroke, myocardial infarction, unstable angina, TIA, symptomatic peripheral vascular disease)
23. History or clinical evidence of thrombo-embolic event
24. History of haemoptysis, cerebral, or clinically significant gastrointestinal haemorrhage in the past 6 months
25. Active bleeding
26. Signs/Suspicion of intestinal obstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Determination of the optimal doses for pazopanib (phase I) | 42 months
Overall response rate according to RECIST criteria / clinical benefit (stable disease or partial response or complete response) (phase II) | 12 weeks after start of treatment

SECONDARY OUTCOMES:
Time to progression (TTP) according to RECIST criteria | 7 years
Overall survival | 7 years
Evaluation of CA125 tumour response | 7 years
Number of patients with Adverse Events | 7 years
Assessment of quality of life over time as defined by EORTC-QLQ C 30 and Ovar 28 questionnaire | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eichbaum, PD Dr. med., Principal Investigator — Medizinische Fakultät Heidelberg Abteilung für Frauenheilkunde und Geburtshilfe
Locations (5):
- Germany (5):
  - Marienkrankenhaus Hamburg, Hamburg
  - Universitäts-Frauenklinik, Heidelberg
  - Klinikum Konstanz Gynäkologie und Geburtshilfe, Konstanz
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz Klinik und Poliklinik für Geburtshilfe und Frauenheilkunde, Mainz
  - Universitätsfrauenklinik Tübingen Klinik für Gynäkologie und Geburtshilfe, Tübingen

REFERENCES:
- [Derived] Dinkic C, Eichbaum M, Schmidt M, Grischke EM, Gebauer G, Fricke HC, Lenz F, Wallwiener M, Marme F, Schneeweiss A, Sohn C, Rom J. Pazopanib (GW786034) and cyclophosphamide in patients with platinum-resistant, recurrent, pre-treated ovarian cancer - Results of the PACOVAR-trial. Gynecol Oncol. 2017 Aug;146(2):279-284. doi: 10.1016/j.ygyno.2017.05.013. Epub 2017 May 19. PMID 28528917
- [Derived] Eichbaum M, Mayer C, Eickhoff R, Bischofs E, Gebauer G, Fehm T, Lenz F, Fricke HC, Solomayer E, Fersis N, Schmidt M, Wallwiener M, Schneeweiss A, Sohn C. The PACOVAR-trial: a phase I/II study of pazopanib (GW786034) and cyclophosphamide in patients with platinum-resistant recurrent, pre-treated ovarian cancer. BMC Cancer. 2011 Oct 20;11:453. doi: 10.1186/1471-2407-11-453. PMID 22014006